CLINICAL TRIAL: NCT06980779
Title: The Correlation of Clinical and Ultrasonographic Findings in Dorsoradial Wrist Pain Patients: Cross Sectional Study
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ilkyazyagar, Medical Doctor, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: E-10840098-202.3.02-3745
Record Dates: First submitted 2025-03-23; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-06

CONDITIONS: Carpometacarpal (CMC) Joint Arthritis; Ganglion Cyst; De Quervain Disease; Radial Neuropathy
Keywords: carpometacarpal joint arthritis; ultrasonography; dorsoradial wrist pain; de Quervain disease; intersection syndrome; ganglion cyst
MeSH Terms: conditions — Capillary Malformations, Congenital, 1; Ganglion Cysts; De Quervain Disease; Radial Neuropathy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: ultrasonographic examination — ultrasonographic examination

SUMMARY:
This study aims to investigate the correlation between ultrasonographic and clinical findings in dorsoradial wrist pain. There are several etiologies for dorsoradial wrist pain, including carpometacarpal joint arthritis, De Quervain's tenosynovitis, proximal and distal intersection syndrome, Wartenberg syndrome, and ganglion cysts. In these clinical scenarios, certain physical examination tests are utilized, such as the Finkelstein test for De Quervain's tenosynovitis; however, this test may also yield positive results in cases of severe joint arthritis. Ultrasonography is proposed as a complementary tool for differential diagnosis. The investigators aim to examine the correlation between clinical test results and ultrasonographic parameters such as tendon thickness in the first extensor compartment, carpometacarpal joint synovitis, cortical irregularities, and the presence of osteophytes. Functional status will be assessed using the QuickDASH and FIHOA questionnaires.

DETAILED DESCRIPTION:
In the assessment of the first carpometacarpal (CMC) joint, the following ultrasonographic parameters will be evaluated: synovitis, presence of osteophytes, joint surface irregularity, and Doppler signal activity. Additionally, conventional hand radiographs of all participants will be reviewed to support the imaging findings.

For the evaluation of De Quervain's tenosynovitis, tendon sheath thickness, tendon cross-sectional area, and intratendinous Doppler activity will be measured. At the anatomical intersection zones of the first dorsal compartment, the presence of peritendinous fluid and associated Doppler activity will also be assessed to identify potential sites of friction or inflammation.

Assessment of the superficial radial nerve will include measurement of its cross-sectional area. A cross-sectional area exceeding one square millimeter will be considered indicative of possible neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* pain in dorsoradial wrist

Exclusion Criteria:

* known rheumatological disease
* history of forearm, wrist, hand fracture
* history of forearm, wrist, hand operation
* mental retardation
* history of major trauma in forearm, wrist and hand
* fibromyalgia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who referred physical theraphy and rehabilitation and orthopedia clinics with dorsoradial wrist and thumb pain
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2024-10-06 (Actual); Study Completion 2024-10-06 (Actual)

PRIMARY OUTCOMES:
Odds Ratio of First Extensor Compartment Tendon Sheath Thickness Associated with De Quervain Disease | At the time of enrollment
  To quantify the association between increased tendon sheath thickness and clinical diagnosis of De Quervain tenosynovitis using logistic regression analysis.
Odds Ratio of Synovial Hypertrophy in CMC Joint Associated with Carpometacarpal Arthritis | At the time of enrollment
  To assess the strength of association between ultrasonographic synovial hypertrophy and clinical diagnosis of carpometacarpal joint arthritis.
Sensitivity of Ultrasonographic Parameters for Diagnosing Dorsoradial Wrist Pathologies | At the time of enrollment
  To assess the diagnostic sensitivity of individual ultrasonographic findings (e.g., tendon sheath thickness, synovial hypertrophy) for detecting De Quervain tenosynovitis and CMC arthritis.
Specificity of Ultrasonographic Parameters for Diagnosing Dorsoradial Wrist Pathologies | At the time of enrollment
  To assess the diagnostic specificity of individual ultrasonographic findings for identifying De Quervain tenosynovitis and CMC arthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Ilkyaz Yağar, Resident, Principal Investigator — University of Health Sciences, FSM Training and Research Hospital, Istanbul; Esra Giray, Associated Professor, Study Director — University of Health Sciences, FSM Training and Research Hospital, Istanbul; Aslınur Keleş, Study Chair — University of Health Sciences, FSM Training and Research Hospital, Istanbul; Feyza Unlu Ozkan, Professor, Study Chair — University of Health Sciences, FSM Training and Research Hospital, Istanbul; Ilknur Aktas, Professor, Study Chair — University of Health Sciences, FSM Training and Research Hospital, Istanbul; Ozge Gulsum Illeez, Associated Professor, Study Chair — University of Health Sciences, FSM Training and Research Hospital, Istanbul
Locations (1):
- University of Health Sciences, FSM Training and Research Hospital, Istanbul, Istanbul, ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McBain B, Rio E, Cook J, Grabinski R, Docking S. Diagnostic accuracy of imaging modalities in the detection of clinically diagnosed de Quervain's syndrome: a systematic review. Skeletal Radiol. 2019 Nov;48(11):1715-1721. doi: 10.1007/s00256-019-03195-z. Epub 2019 Mar 19. PMID 30888457
- [Background] Montechiarello S, Miozzi F, D'Ambrosio I, Giovagnorio F. The intersection syndrome: Ultrasound findings and their diagnostic value. J Ultrasound. 2010 Jun;13(2):70-3. doi: 10.1016/j.jus.2010.07.009. Epub 2010 Sep 19. PMID 23396515
- [Background] Look N, Mcnulty M, Rodriguez-Fontan F, Fenoglio AK. Radial-sided wrist pain differentials: presentation, pathoanatomy, diagnosis, and management. Medicina (B Aires). 2023;83(1):96-107. PMID 36774602